CLINICAL TRIAL: NCT07087587
Title: Sleep Apnea Triggers of Atrial Fibrillation: N-of-1 Randomized Control Trial (SPARTA):
Acronym: SPARTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Mina Chung, MD, Staff of Cardiovascular Medicine, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-548
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Afib; Sleep Apnea Syndrome, Obstructive; CPAP
Keywords: OSA; CPAP; AFIB
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: N of 1 Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alternating CPAP vs. No Treatment (Experimental): Each participant undergoes alternating 2-week periods of CPAP treatment and no treatment over approximately 13 weeks. This personalized intervention evaluates changes in AF burden and quality of life, with patients serving as their own controls.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP will be randomized 2 weeks on 2 weeks off for 12 weeks total

SUMMARY:
A pilot N-of-1 randomized controlled trial evaluating the effectiveness of a personalized CPAP intervention in reducing atrial fibrillation (AF) burden and improving AF-related quality of life in patients with moderate to severe obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
This pilot study investigates whether continuous positive airway pressure (CPAP) therapy reduces AF burden in patients with paroxysmal AF and moderate to severe OSA. Using an N-of-1 randomized crossover design, each participant undergoes alternating 2-week periods with and without CPAP over 3 months. Data on AF episodes are collected from implantable cardiac devices, and AF-related quality of life is assessed using the AFEQT questionnaire. The study also examines CPAP adherence and its correlation with changes in AF burden. Results will inform the design of a larger trial and address gaps in current evidence on the cardiovascular effects of sleep apnea therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Age 18-85 years
3. High burden paroxysmal AF (≥1%)
4. Moderate-severe OSA (AHI ≥ 15)
5. Implanted device with atrial diagnostics
6. Enrolled in remote monitoring

Exclusion Criteria:

1. AF ablation <6 months
2. Valvular abnormalities
3. Excessive daytime sleepiness in safety-critical jobs
4. Plans for ablation during study
5. Non-CPAP OSA treatment
6. Recent device implantation (<6 months)
7. Central sleep apnea

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Average Daily AF Burden (%) | Up to 13 weeks (duration of each patient's participation)
  Percentage change in average daily atrial fibrillation burden, measured via implantable device data, comparing CPAP and non-CPAP periods.

SECONDARY OUTCOMES:
Change in Atrial Fibrillation-Related Quality of Life (AFEQT Score) | Baseline, week 4, week 8, and final visit (~13 weeks)
  Change in patient-reported AFEQT scores between CPAP and non-CPAP periods to assess quality-of-life impact.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehra R, Chung MK, Olshansky B, Dobrev D, Jackson CL, Kundel V, Linz D, Redeker NS, Redline S, Sanders P, Somers VK; American Heart Association Electrocardiography and Arrhythmias Committee of the Council on Clinical Cardiology; and Stroke Council. Sleep-Disordered Breathing and Cardiac Arrhythmias in Adults: Mechanistic Insights and Clinical Implications: A Scientific Statement From the American Heart Association. Circulation. 2022 Aug 30;146(9):e119-e136. doi: 10.1161/CIR.0000000000001082. Epub 2022 Aug 1. PMID 35912643
- [Background] Traaen GM, Aakeroy L, Hunt TE, Overland B, Bendz C, Sande LO, Aakhus S, Fagerland MW, Steinshamn S, Anfinsen OG, Massey RJ, Broch K, Ueland T, Akre H, Loennechen JP, Gullestad L. Effect of Continuous Positive Airway Pressure on Arrhythmia in Atrial Fibrillation and Sleep Apnea: A Randomized Controlled Trial. Am J Respir Crit Care Med. 2021 Sep 1;204(5):573-582. doi: 10.1164/rccm.202011-4133OC. PMID 33938787
- [Background] Caples SM, Mansukhani MP, Friedman PA, Somers VK. The impact of continuous positive airway pressure treatment on the recurrence of atrial fibrillation post cardioversion: A randomized controlled trial. Int J Cardiol. 2019 Mar 1;278:133-136. doi: 10.1016/j.ijcard.2018.11.100. Epub 2018 Nov 20. PMID 30522886
- [Background] Kanagala R, Murali NS, Friedman PA, Ammash NM, Gersh BJ, Ballman KV, Shamsuzzaman AS, Somers VK. Obstructive sleep apnea and the recurrence of atrial fibrillation. Circulation. 2003 May 27;107(20):2589-94. doi: 10.1161/01.CIR.0000068337.25994.21. Epub 2003 May 12. PMID 12743002
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334